CLINICAL TRIAL: NCT04623125
Title: Spaced Retrieval as Treatment for Aphasia: Does Adaptive Spacing Enhance Picture Naming Performance?
Brief Title: Spaced Retrieval as Treatment for Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rotman Research Institute at Baycrest (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Jed A. Meltzer, Ph.D, Senior Scientist, Rotman Research Institute at Baycrest
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-43s
Record Dates: First submitted 2020-10-29; First posted 2020-11-10 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Aphasia, Acquired; Aphasia Primary Progressive
Keywords: Adaptive Spaced-Retrieval; Aphasia; Anomia; Anki
MeSH Terms: conditions — Aphasia; Pick Disease of the Brain; Anomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spaced Repetition (Experimental): Two weeks (10 sessions) of online picture-naming training with 60 words.
  Interventions: Behavioral: Spaced Retrieval Practice

INTERVENTIONS:
Behavioral: Spaced Retrieval Practice — Online picture-naming training with 60 words which the participant experiences word-retrieval difficulties. Cards are shuffled arranged by the computerized training program.

SUMMARY:
Spaced Repetition training has been found to be more effective than massed repetition for individuals with aphasia. This study seeks to examine the relative efficiency of three kinds of spacing for picture-naming training: traditional random presentation, non-adaptive spaced repetition, and adaptive spaced repetition.

DETAILED DESCRIPTION:
Participants undergo a screening evaluation including the Quick Aphasia Battery (administered via teleconferencing software), and a preliminary picture naming test of approximately 300 pictures, used to select individual items for treatment. Participants then undertake online picture naming training for 30 minutes a day, over two weeks. Pictures are repeated according to three different schedules to be compared: random presentation, non-adaptive spaced repetition, and adaptive spaced repetition. We compare the number of pictures successfully learned and the verbal reaction time for the pictures assigned to the three conditions.

ELIGIBILITY:
Inclusion Criteria:

* presence of a post-stroke word finding deficit (i.e. aphasia), or primary progressive aphasia.
* ability to evaluate the correctness of one's own responses when subsequently provided the with the correct answer

Exclusion Criteria:

* diagnosis of a neurological disorder other than post-stroke or primary progressive aphasia
* inability to evaluate the correctness of ones responses when subsequently provided with the correct answer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Picture Naming performance across conditions | Change from baseline to post-intervention immediately after two weeks of daily sessions, and one month followup.
  Word retention assessed after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Baycrest Health Sciences, Toronto, Ontario, Canada